CLINICAL TRIAL: NCT01397890
Title: A Randomised, Parallel-group, Open-label, Multicentre, 3-month Phase IV, Efficacy and Tolerability Study of Budesonide/Formoterol (Symbicort® Turbuhaler® 160/4.5μg/Inhalation, 2 Inhalations Twice Daily) Added to Tiotropium (SpirivaTM 18 μg/Inhalation, 1 Inhalation Once Daily) Compared With Tiotropium (SpirivaTM18 μg/Inhalation, 1 Inhalation Once Daily) Alone in Severe Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Efficacy and Tolerability of Symbicort as an add-on Treatment to Spiriva Compare With Spiriva Alone in Patients With Severe Chronic Obstructive Pulmonary Disease (COPD)
Acronym: SECURE 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D589BL00023
Record Dates: First submitted 2011-06-27; First posted 2011-07-20 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Severe chronic obstructive pulmonary disease (COPD) patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Formoterol Fumarate; Tiotropium Bromide

ARMS (2):
- 1 (Other): Add-on treatment
  Interventions: Drug: Budesonide/formoterol (Symbicort® Turbuhaler®); Drug: Tiotropium (SpirivaTM)
- 2 (Other): Add-on treatment
  Interventions: Drug: Tiotropium (SpirivaTM)

INTERVENTIONS:
Drug: Budesonide/formoterol (Symbicort® Turbuhaler®) — Budesonide/formoterol (Symbicort® Turbuhaler®) 160/4.5μg/inhalation, 2 inhalations twice daily
  Arms: 1
Drug: Tiotropium (SpirivaTM) — Tiotropium (SpirivaTM) 18 μg/inhalation, 1 inhalation once daily

SUMMARY:
This is a multicentre study with a randomised, parallel group, open-label, 3-month phase IV design to assess the efficacy and tolerability of Symbicort as an add-on treatment to Spiriva compare with Spiriva alone in patients with severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Men or women patients ≥40 years of age
* Diagnosis of COPD with symptoms for more than 2 years and there is a history of at least one COPD exacerbation requiring a course of oral steroids and/or antibiotics within 1-12 months before Visit 2
* Forced Expiratory Volume in 1 second (FEV1) ≤50% of predicted normal value, pre-bronchodilator and Forced Expiratory Volume in 1 second (FEV1) / Forced Vital Capacity (FVC) < 70%, pre-bronchodilator
* Total symptom score of 2 or more per day for at least half of run-in period (breathing, cough and sputum scores from the diary card) and complete morning recordings of Digital Peak Flow Meter data at least 7 out of the last 10 days of the run-in period

Exclusion Criteria:

* A history of asthma and seasonal allergic rhinitis before 40 years of age
* Patients who have experienced exacerbation of COPD requiring hospitalisation and /or emergency room treatment and/or a course of oral steroids and/or intravenous corticosteroids and/or antibiotics within 4 weeks prior to Visit 2 and/or during run-in period and also the patients who use of systemic glucocorticosteroids (GCS) within 4 weeks and/or inhaled GCS within 2 weeks prior to Visit 2 and/or during run-in period
* Patients with relevant cardiovascular disorder judged by the investigator
* Patients with glaucoma, prostatic hyperplasia or bladder-neck obstruction judged by the investigator
* Women who are pregnant, breast-feeding or of child-bearing potential judged by the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Chen, M.D., Study Chair — AstraZeneca Pharmaceutical Co., Ltd., Shanghai, China
Locations (31):
- China (8):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Changsha, Hunan
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Guangzhou
- Hong Kong (3):
  - Research Site, Kowloon, HK
  - Research Site, Hong Kong, Hong Kong
  - Research Site, Hong Kong
- Indonesia (3):
  - Research Site, Jakarta
  - Research Site, Solo
  - Research Site, Surabaya
- South Korea (8):
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Jinju, Gyeongsangnam-do
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seoul
- Thailand (9):
  - Research Site, Muang, Changwat Nan
  - Research Site, Nonthaburi, Changwat Nonthaburi
  - Research Site, Chiang Mai, Thailand
  - Research Site, Bangkok
  - Research Site, Chon Buri
  - Research Site, Khon Kaen
  - Research Site, Phitsanulok
  - Research Site, Songkhla
  - Research Site, Udon Thani

REFERENCES:
- [Derived] Lee SD, Xie CM, Yunus F, Itoh Y, Ling X, Yu WC, Kiatboonsri S. Efficacy and tolerability of budesonide/formoterol added to tiotropium compared with tiotropium alone in patients with severe or very severe COPD: A randomized, multicentre study in East Asia. Respirology. 2016 Jan;21(1):119-27. doi: 10.1111/resp.12646. Epub 2015 Sep 23. PMID 26394882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There are 793 patients enrolled. 578 patients were randomized, where there are 287 patients randomized in Symbicort+ Spiriva group and 291 in Spiriva group
Groups:
- Symbicort+Spiriva: Budesonide/formoterol (Symbicort Turbuhaler 160/4.5μg/inhalation, 2 inhalations twice daily) added to tiotropium (Spiriva 18 μg/inhalation, 1 inhalation once daily)
- Spiriva: Spiriva 18 μg/inhalation, 1 inhalation once daily
Period: Overall Study
Arm/Group | Symbicort+Spiriva | Spiriva
Started | 287 | 291
Post-baseline Efficacy Data Collected | 287 ('Full Analysis Set' used for efficacy analysis) | 290 ('Full Analysis Set' used for efficacy analysis)
Received Correct Randomized Treatment | 286 ('Safety Analysis Set' =287+3-1=289. 3 and 1 pts in respective groups received opposite treatment.) | 287 ('Safety Analysis Set' =291+1-3=289.)
Completed | 264 | 260
Not Completed | 23 | 31
Not completed — Withdrawal by Subject | 7 | 11
Not completed — Eligibility Criteria Not Fulfilled | 7 | 6
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 1 | 4
Not completed — Condition under Investigation Worsened | 1 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Severe Non-Compliance to Protocol | 2 | 1
Not completed — Others | 2 | 1

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants is not different from the Milestones.
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort+Spiriva | Spiriva | Total
Number analyzed (Participants) | 287 | 290 | 577
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (7.99) | 66.9 (8.50) | 66.8 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 279 | 273 | 552

OUTCOME MEASURES:

1. Primary Outcome: Pre-dose FEV1
Description: Ratio of pre-dose FEV1 (Forced Expiratory Volume in 1 second) in treatment period to baseline value
Time Frame: Baseline (week 0) and mean in treatment period (weeks 1, 6, 12) measured before inhalation of study drug
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 284 | 277
Ratio | 1.050 [1.030 to 1.070] | 1.006 [0.987 to 1.025]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0004, ANCOVA; multiplicative ANCOVA model with treatment and country as fixed factors and baseline value as a (log-transformed) covariate; Ratio = 1.044, 95% CI 2-sided [1.019 to 1.069]

2. Secondary Outcome: Post-dose FEV1 at 5 Minutes
Description: Ratio of post-dose FEV1 at 5 minutes to baseline value
Time Frame: Baseline (-2 weeks) and mean in treatment period (1, 6, 12 weeks) measured at 5 minutes after inhalation of study drug
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 287 | 286
Ratio | 1.128 [1.109 to 1.147] | 1.045 [1.028 to 1.062]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; Multiplicative ANCOVA model with treatment and country as fixed factors and week 0 pre-dose value as a (log-transformed) covariate; Ratio = 1.079, 95% CI 2-sided [1.057 to 1.102]

3. Secondary Outcome: Post-dose FEV1 at 60 Minutes
Description: Ratio of post-dose FEV1 at 60 minutes to baseline value
Time Frame: Baseline (measured before inhalation of study drug at week 0) and mean in treatment period (measured at 1 hour after inhalation of study drug at weeks 0, 1, 6, 12)
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 287 | 286
Ratio | 1.164 [1.144 to 1.185] | 1.072 [1.053 to 1.091]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Ratio = 1.086, 95% CI 2-sided [1.062 to 1.111]

4. Secondary Outcome: Pre-dose FVC
Description: Ratio of pre-dose FVC (Forced Vital Capacity) in treatment period to baseline value
Time Frame: as for outcome 3
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 284 | 277
Ratio | 1.032 [1.017 to 1.047] | 1.013 [0.999 to 1.029]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0570, ANCOVA; [statistical method as in outcome 2, analysis 1]; Ratio = 1.018, 95% CI 2-sided [0.999 to 1.037]

5. Secondary Outcome: Post-dose FVC at 5 Minutes
Description: Ratio of post-dose FVC at 5 minutes to baseline value
Time Frame: Baseline (measured before inhalation of study drug at week 0) and mean in treatment period (measured at 5 minutes after inhalation of study drug at weeks 0, 1, 6, 12)
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 287 | 286
Ratio | 1.096 [1.081 to 1.110] | 1.044 [1.030 to 1.057]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Ratio = 1.050, 95% CI 2-sided [1.033 to 1.067]

6. Secondary Outcome: Post-dose FVC at 60 Minutes
Description: Ratio of post-dose FVC at 60 minutes to baseline value
Time Frame: as for outcome 3
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 287 | 286
Ratio | 1.116 [1.100 to 1.132] | 1.059 [1.044 to 1.074]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Ratio = 1.054, 95% CI 2-sided [1.036 to 1.073]

7. Secondary Outcome: Pre-dose IC
Description: Ratio of pre-dose IC (Inspiratory Capacity) in treatment period to baseline value
Time Frame: Baseline (week 0) and mean in treatment period (weeks 1, 6, 12) measured before inhalation of study drug
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 265 | 263
Ratio | 1.042 [1.017 to 1.068] | 1.022 [0.998 to 1.047]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.1956, ANCOVA; [statistical method as in outcome 2, analysis 1]; Ratio = 1.020, 95% CI 2-sided [0.990 to 1.050]

8. Secondary Outcome: Post-dose IC at 60 Minutes
Description: Ratio of post-dose IC at 60 minutes to baseline value
Time Frame: as for outcome 3
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 263 | 270
Ratio | 1.154 [1.129 to 1.180] | 1.087 [1.064 to 1.110]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Ratio = 1.062, 95% CI 2-sided [1.035 to 1.091]

9. Secondary Outcome: Pre-dose PEF in Last Week of Treatment
Description: Change in pre-dose morning PEF (Peak Expiratory Flow) from run-in period to last week of treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured before inhalation of study drug in the last week of treatment, up to 12 weeks
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 217 | 208
L/min | 15.753 [7.306 to 24.200] | -4.550 [-13.154 to 4.054]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0001, ANCOVA; Additive ANCOVA model with treatment and centre as fixed factors and the run-in mean of pre-dose morning PEF as a covariate; Mean Difference (Net) = 20.303, 95% CI 2-sided [9.904 to 30.702]

10. Secondary Outcome: Pre-dose PEF in First Week of Treatment
Description: Change in pre-dose morning PEF (Peak Expiratory Flow) from run-in period to first week of treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured before inhalation of study drug in the first week of treatment
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 239 | 241
L/min | 13.405 [8.464 to 18.345] | -0.182 [-4.994 to 4.630]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 13.587, 95% CI 2-sided [7.407 to 19.766]

11. Secondary Outcome: Pre-dose PEF in Whole Treatment Period
Description: Change in pre-dose morning PEF from run-in period to whole treatment period
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured before inhalation of study drug in whole treatment period of 12 weeks
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 256 | 262
L/min | 12.271 [6.382 to 18.160] | -5.198 [-10.925 to 0.530]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 17.469, 95% CI 2-sided [10.147 to 24.791]

12. Secondary Outcome: Post-dose PEF in Last Week of Treatment
Description: Change in post-dose morning PEF at 5 minutes from run-period to last week of treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured at 5 minutes after inhalation of study drug in the last week of treatment, up to 12 weeks
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 177 | 162
L/min | 23.379 [13.199 to 33.560] | -3.049 [-13.556 to 7.458]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 26.428, 95% CI 2-sided [13.463 to 39.393]

13. Secondary Outcome: Post-dose PEF in First Week of Treatment
Description: Change in post-dose morning PEF at 5 minutes from run-in period to first week of treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured at 5 minutes after inhalation of study drug in the first week of treatment
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 186 | 201
L/min | 17.412 [9.349 to 25.476] | 0.220 [-7.486 to 7.926]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0006, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 17.192, 95% CI 2-sided [7.491 to 26.894]

14. Secondary Outcome: Post-dose PEF in Whole Treatment Period
Description: Change in post-dose morning PEF at 5 minutes from run-period to whole treatment period
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured at 5 minutes after inhalation of study drug in whole treatment period of 12 weeks
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 248 | 247
L/min | 15.880 [9.307 to 22.454] | -2.591 [-9.063 to 3.880]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 18.472, 95% CI 2-sided [10.347 to 26.596]

15. Secondary Outcome: Use of Reliever Medication During Day in the Last Week on Treatment
Description: Change in the number of inhalations of reliever medication during day from run-in period to the last week on treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured during day in the last week on treatment, up to 12 weeks
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 274 | 274
times/day | -0.750 [-0.935 to 0.566] | -0.082 [-0.267 to 0.103]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.668, 95% CI 2-sided [-0.900 to -0.437]

16. Secondary Outcome: Use of Reliever Medication During Day in the First Week on Treatment
Description: Change in the number of inhalations of reliever medication during day from run-in period to the first week on treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured during day in the first week on treatment
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 284 | 284
times/day | -0.457 [-0.598 to -0.316] | -0.082 [-0.222 to 0.058]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.375, 95% CI 2-sided [-0.552 to -0.198]

17. Secondary Outcome: Use of Reliever Medication During Day in the Whole Treatment Period
Description: Change in the number of inhalations of reliever medication during day from run-in period to the whole treatment period
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured during day in the whole treatment period of 12 weeks
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 284 | 286
times/day | -0.685 [-0.836 to -0.533] | -0.134 [-0.284 to 0.016]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.551, 95% CI 2-sided [-0.741 to -0.361]

18. Secondary Outcome: Use of Reliever Medication During Night in the Last Week on Treatment
Description: Change in the number of inhalations of reliever medication during night from run-in period to the last week on treatment
Time Frame: as for outcome 15
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 272 | 275
times/day | -0.174 [-0.299 to -0.049] | 0.062 [-0.062 to 0.187]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0028, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.236, 95% CI 2-sided [-0.391 to -0.082]

19. Secondary Outcome: Use of Reliever Medication During Night in the First Week on Treatment
Description: Change in the number of inhalations of reliever medication during day from run-in period to the first week on treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured during night in the first week on treatment
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 283 | 286
times/day | -0.113 [-0.206 to -0.019] | 0.011 [-0.081 to 0.104]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0372, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.124, 95% CI 2-sided [-0.240 to -0.007]

20. Secondary Outcome: Use of Reliever Medication During Night in the Whole Treatment Period
Description: Change in the number of inhalations of reliever medication during night from run-in period to the whole treatment period
Time Frame: as for outcome 17
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 285 | 286
times/day | -0.241 [-0.336 to -0.147] | -0.010 [-0.104 to 0.084]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.231, 95% CI 2-sided [-0.350 to -0.113]

21. Secondary Outcome: Change in COPD Symptoms - Breathing
Description: Change in breathing symptom score (from 0:none to 4:severe) from run-in period
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements in the whole treatment period of 12 weeks
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 284 | 286
score on a scale | -0.372 [-0.454 to -0.290] | -0.110 [-0.191 to -0.029]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.262, 95% CI 2-sided [-0.364 to -0.159]

22. Secondary Outcome: Change in COPD Symptoms - Cough
Description: Change in Cough symptom score (from 0:none to 4:severe) from run-in period
Time Frame: as for outcome 21
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 283 | 286
score on a scale | -0.311 [-0.394 to -0.229] | -0.169 [-0.250 to -0.087]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0067, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.143, 95% CI 2-sided [-0.246 to -0.040]

23. Secondary Outcome: Change in COPD Symptoms - Sputum
Description: Change in Sputum symptom score (from 0:none to 4:severe) from run-in period
Time Frame: as for outcome 21
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 284 | 286
score on a scale | -0.216 [-0.295 to -0.136] | -0.094 [-0.173 to -0.014]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0171, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = -0.122, 95% CI 2-sided [-0.222 to -0.022]

24. Secondary Outcome: COPD Exacerbations
Description: Severe exacerbations requiring systemic steroids (oral ≥3 days or parenteral) or hospitalisation or emergency room treatment due to worsening of COPD symptoms
Time Frame: Whole treatment period of 12 weeks
Population: FAS (287 + 290); less number of patients analyzed was caused by missing values.
Measure: Least Squares Mean (95% Confidence Interval); unit: exacerbations/participant/12 weeks
Arm/Group | Symbicort+Spiriva | Spiriva
Number analyzed (Participants) | 287 | 290
exacerbations/participant/12 weeks | 0.182 [0.138 to 0.239] | 0.307 [0.248 to 0.379]
Statistical Analysis 1: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0032, Poisson regression; Poisson regression model with treatment as a factor and the duration time in study as an offset variable morning PEF as a covariate; Rate ratio = 0.593, 95% CI 2-sided [0.419 to 0.839]
Statistical Analysis 2: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0167, Regression, Cox; Time to the first COPD exacerbation; Cox Proportional Hazard = 0.614, 95% CI 2-sided [0.412 to 0.916]
Statistical Analysis 3: Comparison: Symbicort+Spiriva vs Spiriva; Test type: Superiority or Other; p = 0.0196, Log Rank

ADVERSE EVENTS:
Time Frame: 12 weeks of treatment period
Arm/Group | Symbicort+Spiriva | Spiriva
Serious Adverse Events (participants affected / at risk) | 14/289 | 24/289
Other Adverse Events (participants affected / at risk) | 75/289 | 76/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symbicort+Spiriva (N=289) | Spiriva (N=289)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (13)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestion (Cardiac disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Bile duct cancer (Hepatobiliary disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Joint dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symbicort+Spiriva (N=289) | Spiriva (N=289)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colon adenoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Post herpetic neuralgia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sputum abnormal (Investigations) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI Disclosure Restriction is indicated in the Clinical Study Agreement, please refer to this document of each PI and country.